CLINICAL TRIAL: NCT02397265
Title: Clinical Assessment of a Closed-loop System With Glucagon, Exercise and Mixed Meals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 14SM2107
Record Dates: First submitted 2015-03-05; First posted 2015-03-24 (Estimated); Results first posted 2019-11-01 (Actual); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 diabetes; Hypoglycaemia; Closed loop insulin pump; Artificial pancreas; Exercise; Mixed meals; Bihormonal pump
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Bihormonal closed loop (Experimental): Bi-hormonal closed loop pump will be used in the exercise and mixed meal substudies
  Interventions: Device: Bi-hormonal closed loop pump
- Standard opened loop pump (Active Comparator): Standard opened loop pump will be used in the exercise and mixed meal substudies
  Interventions: Device: Standard opened loop pump
- Insulin only (Placebo Comparator): Insulin only closed loop
  Interventions: Device: Insulin closed loop

INTERVENTIONS:
Device: Bi-hormonal closed loop pump — Using a bio-inspired artificial pancreas consisting of a bi-hormonal closed loop pump
  Arms: Bihormonal closed loop
Device: Standard opened loop pump — Using a standard opened loop pump
  Arms: Standard opened loop pump
Device: Insulin closed loop — Using a closed loop
  Arms: Insulin only

SUMMARY:
The diabetes technology group at Imperial College have developed a bio-inspired artificial pancreas (BiAP) system which uses a control algorithm based on a mathematical model of beta-cell physiology. The algorithm is implemented on a miniature silicon microchip within a portable handheld device, which interfaces the components of the artificial pancreas.

Development of closed-loop insulin delivery devices to intensify control without hypoglycaemia has been extensively reviewed and have shown encouraging results . However, they have not yet proven to be robust when challenged with uncertainty and the external challenges (such as mixed meal contents, physical exercise, physiological stress and intercurrent illness) that people with Type 1 Diabetes Mellitus (T1DM) may be exposed to outside the clinical environment.

The principal research objective is to assess the safety and efficacy of a closed-loop system for T1DM compared to standard insulin pump therapy (open-loop). The primary outcome from the studies will be % time spent with a glucose concentration in the target range (3.9-10.0mmol/l). This outcome incorporates safety as it ensures subjects do not have low or high glucose excursions and is the principal measure of efficacy for closed-loop insulin delivery systems in the scientific literature. Other measured outcomes will be % time spent in euglycaemia (3.9-7.8mmol/l), % time spent in hypoglycaemia (<3.9mmol/l), % time spent in hyperglycaemia (>10mmol/l), mean venous blood and sensor glucose, glycaemic variability as measured by standard metrics (Standard Deviation, Continuous Overlapping Net Glycaemic Action, Lability Index, J-Index, Glycaemic Risk Assessment Diabetes Equation, Mean Of Daily Differences, Mean Amplitude of Glucose Excursion, Average Daily Risk Range, M-VALUE, Mean Average Glucose), glycaemic risk as measured by Low Blood Glucose Index (LBGI) and High Blood Glucose Index (HBGI), closed-loop error grid analysis, glucose area under the curve. All measures have been previously published and validated.

This clinical trial protocol assesses the artificial pancreas system in three separate sub-studies:

1. In a bi-hormonal (insulin and glucagon) configuration
2. During and after exercise with bi-hormonal closed loop, and standard insulin opened loop
3. During and after meals of mixed composition with bi-hormonal closed loop, and standard insulin opened loop

DETAILED DESCRIPTION:
Methodology Randomised controlled cross-over open label study

Sub study 1 (n=10)

In sub-study 1 which includes the first bio-inspired artificial pancreas study using bi-hormonal (insulin and glucagon) control a fasting 6-hour bi-hormonal closed-loop study will be conducted to assess proof of concept and safety prior to the 25-hour randomised controlled crossover study

Each subject will then be randomised to attend either a closed-loop visit or an open-loop visit first. Once either visit is completed each subject will crossover and attend the remaining visit.

Sub-study 2 (n=20) The aim of sub-study 2 is to challenge the bi-hormonal pump during a moderate exercise. Subjects will be initially randomised to either the bi-hormonal or the standard opened loop and then cross over. Each study will last for 25 hours

• Exercise protocol: Subjects will be connected to the gas analyser and heart rate/ECG monitor as per COSMED manufacturer instructions.

The oxygen consumption (VO2)/Carbon dioxide production (VCO2) and heart rate/ECG trace will be displayed continuously in real time while the subject is exercising.

Warm-up: 3 minutes of cycling at low resistance (20-30 watts) while maintaining a speed of 60-80 revolutions per minute After the warm-up the subjects will undergo a 30 minutes moderate intensity exercise session on the bike aiming to maintain their VO2 between 10-20% above their 1st ventilatory anaerobic threshold. If their VO2 falls below or goes above this level then the resistance will be increased or decreased accordingly. The target VO2 and the starting resistance (watts) will be individually set based on their baseline exercise test outcome.

The estimated time needed to complete the exercise test is 35-40 minutes.

Real-time continuous glucose monitoring alarms will be set at 4mmol/L and 15mmol/L and will be audible by the subject and the research team.

The glucagon solution will be replaced with a freshly reconstituted glucagon solution every 8 hours throughout the closed-loop study If the venous blood glucose concentrations fall below 3.5mmol/L or if the subject experiences hypoglycaemia symptoms then hypoglycaemia will be confirmed by an additional venous blood plasma glucose sample and will be treated according to Imperial College Hospitals National Health Service Trust Guidelines.

After 25 hours of closed-loop, at 12:00 the next day, the subject's own insulin pump will be primed, reconnected and started as per the subject's usual insulin regime. Once running, the closed loop system will be disconnected. The subject can then eat and drink freely and may be discharged after 2 hours, or when glucose concentrations are stable.

The same protocol will be used when subjects cross over for the standard opened loop 25 hour study for the remaining visit.

Sub-study 3: Bi-hormonal closed-loop control during- and after mixed meals (n=20) A high fat/high carbohydrate content dinner (45g fat, 80g CHO) will be given at 19:00, a high glycaemic index breakfast (40g CHO) at 07:00 and a high protein/low carbohydrate lunch ( 30g protein,10g CHO) at 12:00.

Subjects will be free to gently mobilise around the clinical research unit, smoking will not be permitted. Subjects may drink unlimited water throughout the visit.

Real-time continuous glucose monitoring alarms will be set at 4mmol/L and 15mmol/L and will be audible by the subject and the research team.

The glucagon solution will be replaced with a freshly reconstituted glucagon solution every 8 hours throughout the closed-loop studies.

If the venous blood glucose concentrations fall below 3.5mmol/L or if the subject experiences hypoglycaemia symptoms then hypoglycaemia will be confirmed by an additional venous blood plasma glucose sample and will be treated according to Imperial College Hospitals National Health Service Trust Guidelines.

After 25 hours of closed-loop, at 18:00 the next day, the subject's own insulin pump will be primed, reconnected and started as per the subject's usual insulin regime. Once running, the closed-loop system will be disconnected. The subject can then eat and drink freely and may be discharged after 2 hours, or when glucose concentrations are stable.

The same protocol will be applied after cross over but with a standard opened loop insulin pump for the remaining visit.

ELIGIBILITY:
Inclusion Criteria:

* Adults over 18 years of age
* Type 1 diabetes confirmed on the basis of clinical features and a fasting c-peptide <200 pmol/L
* Type 1 diabetes for greater than 1 year
* Continuous subcutaneous insulin infusion for greater than 6 months
* HbA1c < 10% (86mmol/mol)

Exclusion Criteria:

* Recurrent severe hypoglycaemia and hypoglycaemia unawareness
* Pregnant or planning pregnancy
* Breastfeeding
* Enrolled in other clinical trials
* Have active malignancy or under investigation for malignancy
* Allergic to lactose
* Allergic to glucagon

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-12-03 (Actual); Primary Completion 2015-07-22 (Actual); Study Completion 2015-07-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nick Oliver, MRCP, Principal Investigator — Imperial College London
Locations (1):
- Imperial College, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nathan D, Cleary P, Backlund J, Genuth S, Lachin J, Orchard T, Raskin R, Zinman B. Diabetes Control and Complications Trial/Epidemiology of Diabetes Interventions and Complications (DCCT/EDIC) Study Research Group. Intensive diabetes treatment and cardiovascular disease in patients with type 1 diabetes,
- [Background] Buckingham B, Wilson DM, Lecher T, Hanas R, Kaiserman K, Cameron F. Duration of nocturnal hypoglycemia before seizures. Diabetes Care. 2008 Nov;31(11):2110-2. doi: 10.2337/dc08-0863. Epub 2008 Aug 11. PMID 18694975
- [Background] Sovik O, Thordarson H. Dead-in-bed syndrome in young diabetic patients. Diabetes Care. 1999 Mar;22 Suppl 2:B40-2. PMID 10097898
- [Background] Hovorka R. Closed-loop insulin delivery: from bench to clinical practice. Nat Rev Endocrinol. 2011 Feb 22;7(7):385-95. doi: 10.1038/nrendo.2011.32. PMID 21343892
- [Background] Cobelli C, Renard E, Kovatchev B. Artificial pancreas: past, present, future. Diabetes. 2011 Nov;60(11):2672-82. doi: 10.2337/db11-0654. No abstract available. PMID 22025773
- [Background] Ward WK, Massoud RG, Szybala CJ, Engle JM, El Youssef J, Carroll JM, Roberts CT Jr, DiMarchi RD. In vitro and in vivo evaluation of native glucagon and glucagon analog (MAR-D28) during aging: lack of cytotoxicity and preservation of hyperglycemic effect. J Diabetes Sci Technol. 2010 Nov 1;4(6):1311-21. doi: 10.1177/193229681000400604. PMID 21129325
- [Background] Oliver N, Georgiou P, Johnston D, Toumazou C. A benchtop closed-loop system controlled by a bio-inspired silicon implementation of the pancreatic beta cell. J Diabetes Sci Technol. 2009 Nov 1;3(6):1419-24. doi: 10.1177/193229680900300623. PMID 20144397
- [Background] Herrero P, Georgiou P, Oliver N, Johnston DG, Toumazou C. A bio-inspired glucose controller based on pancreatic beta-cell physiology. J Diabetes Sci Technol. 2012 May 1;6(3):606-16. doi: 10.1177/193229681200600316. PMID 22768892
- [Background] Herrero P, Georgiou P, Oliver N, Reddy M, Johnston D, Toumazou C. A composite model of glucagon-glucose dynamics for in silico testing of bihormonal glucose controllers. J Diabetes Sci Technol. 2013 Jul 1;7(4):941-51. doi: 10.1177/193229681300700416. PMID 23911175

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 24 participants were recruited (due to 4 withdrawals before randomization) to reach a total n=20 for the study. Only 6 were randomised/completed due to sufficient data, rest of 14 people did not do the study. 6 people were randomized and completed the study for each arm. The interventions were in random order according to the randomisation.
Groups:
- First Bihormonal Closed Loop: Bihormonal Closed Loop first, then Standard Opened Loop Pump, then Insulin
- First Standard Opened Loop Pump: First Standard Opened Loop Pump, then Bihormonal Closed Loop, then Insulin
- First Insulin Only: First Insulin, then Standard Opened Loop Pump, then Bihormonal Closed Loop
Period: First Intervention of Three
Arm/Group | First Bihormonal Closed Loop | First Standard Opened Loop Pump | First Insulin Only
Started | 2 | 2 | 2
Completed | 2 | 2 | 2
Not Completed | 0 | 0 | 0
Period: Second Intervention of Three
Arm/Group | First Bihormonal Closed Loop | First Standard Opened Loop Pump | First Insulin Only
Started | 2 | 2 | 2
Completed | 2 | 2 | 2
Not Completed | 0 | 0 | 0
Period: Third Intervention of Three
Arm/Group | First Bihormonal Closed Loop | First Standard Opened Loop Pump | First Insulin Only
Started | 2 | 2 | 2
Completed | 2 | 2 | 2
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participant: Crossover study, all participant
Arm/Group | All Participant
Number analyzed (Participants) | 6
Age, Continuous [Mean (Full Range); unit: years] | 55 [50 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 2
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 6

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Time in Target Range Over 24 Hour
Description: The primary outcome from the studies will be time spent with a glucose concentration in the target range (3.9-10.0mmol/l).
Time Frame: 24 hours
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | Bihormonal Closed Loop | Standard Opened Loop Pump | Insulin Only
Number analyzed (Participants) | 6 | 6 | 6
percentage of time | 2 [0.4 to 3] | 4.7 [1.8 to 12] | 1.3 [0.4 to 7.2]

ADVERSE EVENTS:
Time Frame: 24 hours
Arm/Group | Bihormonal Closed Loop | Standard Opened Loop Pump | Insulin Only
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes